CLINICAL TRIAL: NCT02022488
Title: Prevention of Emergence Agitation in Children After Sevoflurane Anesthesia With Ketamine-midazolam Combination: A Prospective Randomized Clinical Trial
Brief Title: Sevoflurane Induced Emergence Agitation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yeditepe University Hospital (Other)
Responsible Party: Principal Investigator, Sevgi Bilgen, Yeditepe University, Yeditepe University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 162
Record Dates: First submitted 2013-12-10; First posted 2013-12-27 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Emergence Agitation
Keywords: Child; Sevoflurane; Emergence delirium; General anesthesia; Premedication.
MeSH Terms: conditions — Emergence Delirium | interventions — Midazolam; Alfentanil; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- midazolam and alfentanil (Active Comparator): Midazolam 0.5mg/kg (oral) Alfentanil 10 microgram/kg (oral)
  Interventions: Drug: midazolam; Drug: alfentanil
- midazolam and ketamine (Active Comparator): Midazolam 0.5mg/kg (oral) Ketamine 2mg/kg (intranasal)
  Interventions: Drug: midazolam; Drug: ketamine
- midazolam (Placebo Comparator): Midazolam 0.5mg/kg
  Interventions: Drug: midazolam

INTERVENTIONS:
Drug: midazolam — Group M
Drug: alfentanil — Group MA
  Arms: midazolam and alfentanil
Drug: ketamine — Group MK
  Arms: midazolam and ketamine

SUMMARY:
Investigators evaluated the effect of intranasal ketamine or alfentanil addition to oral midazolam for prevention of emergence agitation.Seventy-eight, 1-8 year-old children, undergoing urological surgery with sevoflurane anesthesia was included in the study. All the children received oral midazolam 0.5 mg/kg 40 minutes before anesthesia induction then enrolled to one of the study groups, randomly. Ketamine group (Group MK; n=26) patients were given 2mg/kg intranasal ketamine whereas, alfentanil group (Group MA; n=25) were given 10microgram/kg intranasal alfentanil 8-10 min before the induction of anesthesia. Saline group (Group MS; n=27) received intranasal isotonic saline.Parental separation, mask acceptance were evaluated with a 4- point scale. Emergence agitation was evaluated with Pediatric Anesthesia Emergence Delirium score.

ELIGIBILITY:
Inclusion Criteria:

* 1- 8 years
* American Society of Anesthesiologist (ASA) I-II,
* Patients undergoing procedures below the umbilicus

Exclusion Criteria:

* cardiac diseases
* pulmonary diseases
* hepatic diseases
* renal diseases
* psychological or emotional disorders

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Pediatric Anesthesia Emergence Delirium (PAED) score | 7 months
  Emergence agitation was evaluated using the Pediatric Anesthesia Emergence Delirium (PAED) score

SECONDARY OUTCOMES:
Parental separation score | 7 months
  Parental separation were evaluated with a 4- point scale in the preoperative period
Mask acceptance | 7 months
  The ease of mask acceptance were evaluated with a 4- point scale in the preoperative period

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University Hospital, Istanbul, Turkey (Türkiye)